CLINICAL TRIAL: NCT00786175
Title: A Cross-sectional Observational Survey to Evaluate the Rate of Diabetes and Glucose Intolerance (Both Diagnosed and Undiagnosed) Among Hong Kong Chinese Subjects With Coronary Heart Disease
Brief Title: A Survey to Evaluate the Rate of Abnormal Glucose Tolerance Among Hong Kong Chinese Subjects With Coronary Heart Disease
Status: Withdrawn | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Juliana Chan, Chair Professor of Medicine and Therapeutics, Chinese University of Hong Kong
Other Study IDs: CRE-2008.336
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Coronary Heart Disease; Diabetes Mellitus
MeSH Terms: conditions — Coronary Disease; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Hypothesis: there is a high prevalence rate of diabetes, including asymptomatic undiagnosed glucose intolerance, among subjects with coronary heart disease in Hong Kong.

A cross-sectional survey is planned to study the rate of undiagnosed diabetes and glucose intolerance among the Chinese patients with coronary heart disease in Hong Kong. The survey results will be important for us to plan the logistics to investigate and manage the potential glucose abnormality of our heart disease patient.

DETAILED DESCRIPTION:
Diabetes is becoming an epidemic in Hong Kong, affecting over 10% of population and causing a major burden to the health care system. Over 30-40% of patients admitted to the medical wards of the Hospital Authority hospitals have diabetes as a contributory factor. It was estimated that thirty to fifty percent of patients with stroke, heart failure or acute myocardial infarction have diabetes as a key causative factor. However, the exact prevalence rate of diabetes, including asymptomatic undiagnosed glucose intolerance, among subjects with coronary heart disease is still unknown in Hong Kong. Many heart disease patients with undiagnosed diabetes remained being untreated on their abnormal glycemic status, which will further aggravate the heart disease and impair the prognosis.

The investigators plan to conduct a cross-sectional survey to study the rate of undiagnosed diabetes and glucose intolerance among the Chinese patients with coronary heart disease in Hong Kong. The survey results will be important for us to plan the logistics to investigate and manage the potential glucose abnormality of our heart disease patient.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years
2. Subjects admitted to Hospital Authority hospital as in-patients (AHNH) with the diagnosis of coronary heart disease (ICD code 410-414) during the period 1 April 2007 to 31 March 2008.
3. Subjects admitted to AHNH for the procedure Percutaneous Coronary Intervention (PCI) to manage coronary heart disease.

Exclusion Criteria:

1. Known Type 1 diabetes defined as history of ketosis [acute symptoms with heavy ketonuria (>3+) or ketoacidosis] or heavy ketonuria (3+) or continuous requirement of insulin treatment within one year of diagnosis and thereafter.
2. Patients with terminal malignancy or other life-threatening diseases with less than 6-month expected survival
3. Patients with a mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hong Kong Chinese with history of coronary heart disease being diagnosed in 2008 in HA hospitals
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-10; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Ko, MD, Principal Investigator — Asia Diabetes Foundation
Locations (1):
- Hong Kong Institute of Diabetes and Obesity, Hong Kong, China